CLINICAL TRIAL: NCT07124208
Title: A Randomized Double-Blinded and Placebo-Controlled Trial to Assess the Efficacy of Biophoton Therapy to Treat Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Institute of All Medicines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIAM-DM2025
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes, Biophotons, Ageing Marker, Stem Cells,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This is a 2-group comparison study. The biostatistician will prepare a randomization schedule including a series of subject numbers. A subject number will be randomly assigned to each study participant, which will assign them to either the control group or the treatment group. This phase lasts for 4 weeks. At the end of Week 4, the active devices will replace the placebo. Both groups will be actively participating in the study for 2 months (8 weeks).
  Other than the Informed Consent Form (ICF), all study information will be recorded using the subject number.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The same shape, size, and weight of the device without generating biophoton is to be labeled with a random code and used as a comparator. The comparator device will be packed and used in the same way as the Treatment devices. Each two units will be packed inside a black container. Each package will be placed on each side of the bed and used during night sleep. The 8 study devices will be used during the entire study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): The same size, shape, and weight of the devices without emitting biophotons will be provided and used during the first 4 weeks of the randomized study period.
  Interventions: Device: Biophoton Generators
- Treatment (Experimental): Eight Tesla Biophotonizer-A will be packed in 4 sleeves and used during the study. The Placebo will be packed the same way without emitting biophotons.
  Interventions: Device: Biophoton Generators

INTERVENTIONS:
Device: Biophoton Generators — Biophoton Generators will be placed around the subject's bed and used during the night sleep during the entire study period.

SUMMARY:
Study Objective The purpose of this clinical study is to evaluate if biophoton therapy, delivered by Tesla BioHealing® Biophoton Generators (Biophotonizer), can treat diabetes.

Study Design This is a randomized, double-blind, placebo-controlled intervention clinical study to assess the effectiveness of biophoton therapy in treating diabetes. Approximately 46 volunteers will participate in the study.

Study Randomization The biostatistician will prepare a randomization schedule including a serial of subject numbers. A subject number will be randomly assigned to each study participant, which will assign them to either the control group or the treatment group. This phase lasts for 4 weeks. At the end of Week 4, the active devices will replace the placebo. Both groups will be actively participating in the study for 2 months (8 weeks).

Other than the Informed Consent Form (ICF), all study information will be recorded by using the subject number.

The Principal Investigator, study physicians, study nurses, data-entry specialists, and biostatisticians, as well as the participants, will be blinded about who received which product during the first two weeks of study participation.

Study Enrollment Each potentially qualified volunteer will review the Informed Consent Form online (e-ICF) and Enrollment Criteria online (e-Criteria) first, then discuss the e-ICF and e-Criteria with the study team medical professional via telephone during the scheduled time. Each qualified volunteer will sign the e-ICF and send it to the Medical Office Coordinator. The study coordinator will assign the qualified volunteer a randomized subject number, then the volunteer will become a study participant.

DETAILED DESCRIPTION:
Study Procedure We expect that participants will remain in this clinical treatment for two months. The first 4 weeks of participation are double-blinded to record the placebo effects, as each set of the study device is labelled with a unique code for use by only one participant. The change of the placebo device to the treatment device will be performed by the study device management team staff, who will not inform the study participant or the study research staff who are involved in study data collection. Each participant assigned to the Control Group will be treated with 8 placebo devices, with two devices placed on the 2 sides of the bed. Each participant assigned to the Treatment Group will receive 8 Biophoton generator Biophotonizer- A devices and placed on the 2 sides of the bed. Each participant will use the Treatment or Control device for at least 8 hours every night for 8 weeks during sleep. During the day, participants are welcome to bring the study devices and place them near their bodies. At the end of the initial 4 weeks, study participants randomized to the Placebo group will be switched to the Open-Label product to treat them for 1 month (4 weeks).

Each participant will be guided by study team staff to perform the following tests on their assigned testing days: the standard SF-36 questionnaires (SF-36) for measuring life quality, and other study indicators, respectively, at the Baseline, bi-weekly after using the study devices.

Study Supply The 8 study devices (Placebo or Treatment) will be packed inside the two specially made black carriers for easy use.

Each participant will use the assigned devices during the first 4-week randomized period. The active devices will be used for 8 weeks, during the active treatment period in the Treatment Group, and 4 weeks in the Control Group.

Study Patient Population An adult who is clinically diagnosed with diabetes mellitus type 2 (DM2) can participate in this clinical trial.

Investigational Product and Mode of Administration Tesla BioHealing Biophotonizer-A is an over-the-counter (OTC) medical device that can be used by anyone who wants to increase blood circulation and reduce bodily pains. For this study, the coded active or inactive Biophotonizer-A will be placed on each side of the bed during overnight sleep for four weeks. Then, all participants will use open-label active devices for 4 weeks, or 8 weeks if in the Treatment Group.

Comparator and Mode of Administration The same shape, size, and weight of the device without generating biophotons is to be labeled with a random code and used as a comparator. The comparator device will be packed and used in the same way as the Treatment devices. Each two units will be packed inside a black container. Each package will be placed on each side of the bed and used during nighttime sleep. The 8 study devices will be used during the entire study period.

Study Duration Estimated date of the first patient enrolled: August 15, 2025. The estimated date of the last participant is August 14, 2026.

Duration of Treatment Participants in the Treatment Group and Control Group will actively participate in the study for 4 weeks during the randomization period. The treatment group will be continually treated for 4 more weeks. The control group will be treated for 4 weeks after the first 4 weeks of placebo observation.

Outcome Variables

Primary Outcome Measure:

Fasting Glucose [Time Frame: baseline, 0-4, and 0-8 weeks].

Secondary Outcome Measure:

1. Sugar Attachment (HbA1c) [Time Frame: baseline, 0-4, and 0-8 weeks]. HbA1C is an indicator of sugar attachment. This indicator will be measured at the baseline, week 4, and week 8.
2. Blood Lipids [Time Frame: baseline, 0-4, and 0-8 weeks]. Blood lipids are indicators of the body's metabolism and cardiologic health. This indicator will be measured at the baseline, weeks 4 and 8.
3. Stem cell counts [Time Frame: baseline, 0-4, and 0-8 weeks]. Stem cells are indicators of the body's regenerative capacity and biological health.
4. Biomarkers of aging [Time Frame: baseline, 0-4, and 0-8 weeks]. Biomarkers of aging are indicators of a person's biological age, which may differ from their chronological age, and reflect the rate of aging, health status, and risk of age-related diseases.
5. Blood Flow Assessment. [Time Frame: baseline, 0-4, and 0-8 weeks]. Blood flow will be evaluated using the Falcon Quad device, a non-invasive and painless diagnostic tool designed to assess vascular function by measuring and comparing blood pressure across different regions of the body. This method provides clinically valuable, real-time insights into systemic and peripheral circulation, helping to monitor vascular health and treatment response in participants with diabetes. The assessment reflects underlying arterial conditions that may be affected by diabetic vascular complications.
6. Blood Pressure. [Time Frame: baseline, 0-2, 0-4, 0-6, and 0-8 weeks]. Blood pressure is an indicator of blood circulation and cardiovascular health. This indicator will be measured at the baseline, week 2, 4, 6, and 8.
7. Body Weight. [Time Frame: baseline, 0-2, 0-4, 0-6, and 0-8 weeks]. Body weight is an indicator of the body's metabolism and overall health. This indicator will be measured at the baseline, weeks 4 and 8.
8. Life Quality. Short Form Health Survey (SF-36) [Time Frame: baseline, 0-2, 0-4, 0-6, and 0-8 weeks] is to measure the quality of life as influenced by the investigational medical device. SF-36 has been used worldwide as a standard clinical research tool.
9. Diabetes Medicine use. The reported use of diabetic medicine will be tabulated and analyzed. [Time Frame: baseline, baseline, 0-2, 0-4, 0-6, and 0-8 weeks].
10. Diabetic Group Symptoms (DGS). [Time Frame: baseline, 0-2, 0-4, 0-6, and 0-8 weeks]. The DGS measures the impact of biophoton therapy on the most common diabetic symptoms and signs using the 10-Leeloc scale. The improved DGS includes:

1) Reduces frequent urination 2) Reduces thirst 3) Reduces hunger 4) Reduced blurred vision 5) Increased mental clarity 6) Increases wound healing speed 7) Reduce stress and anxiety 8) Improve social activities 9) Reduces inflammation 10) Reduces pain from diabetes 11) Reduces fatigue 12) Promotes restful sleep 13) Improved memory 14) Increases physical strength 15) Enhances sexual function 16) Reduces the frequency of infections 17) Reduces tingling in hands or feet 18) Reduces peripheral neuropathy Safety Outcome: Occurrence of adverse events. Any adverse events were reported by participants. [Time Frame: Any Adverse Events occurred at the baseline, and up to 8 weeks.] Any adverse events reported by participants will be tabulated and compared between the two groups.

Eligibility Criteria

Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Is able and willing to comply with all trial requirements.
* Male or female aged 18-70 years old without major diseases.
* An adult clinically diagnosed with DM2
* Participants must not be heavy users of Tesla BioHealing devices; enrollment will be determined by the clinical team based on an evaluation of the participant's prior device usage.
* Must be fluent in English.

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by research medical professionals.
* Is participating in another investigational drug or device trial Statistical Methods The sample size is calculated based on the primary efficacy variable and the data from the pilot study in diabetes patients (more than 70% success for the treatment, and less than 10% success for the Placebo) to compare the treatment with the Biophoton Generator, which was at least 70% successful, and to compare with the placebo.

The treatment success is defined as a 50% efficacy in lowering fasting glucose during the first two-week study period. To be conservative, one successful rate, 50% for the Treatment, 20% for the Control was used to calculate sample sizes, see table below.

Possibility Number Control Success Rate % Treatment Success Rate* % Power Confidence Level Sample Size per Group Additional 20% per Group 1 20% 50% 90% 95% 19 4

*Treatment success is defined as the fasting glucose becoming normal in at least 50% study participants as compared to Baseline.

We plan to enroll 23 Participants in each group to have 19 completers by adding 4 (20%) more participants. Therefore, a total of 46 participants will be enrolled. If the Principal Investigator decides to increase the enrollment to enable a statistical difference between the two groups, the enrollment can continue. Primary and secondary outcome variables will be statistically analyzed by using Chi-square analysis or paired T-test.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial.
* Is able and willing to comply with all trial requirements.
* Male or female aged 18-70 years old without major diseases.
* An adult clinically diagnosed with DM2
* Participants must not be heavy users of Tesla BioHealing devices; enrollment will be determined by the clinical team based on an evaluation of the participant's prior device usage.
* Must be fluent in English.

Exclusion Criteria:

* Untreated psychiatric disturbances that would affect trial participation as judged by research medical professionals.
* Is participating in another investigational drug or device trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Fasting Glucose | [Time Frame: baseline, 0-4, and 0-8 weeks]
  Fasting Glucose at Baseline, Week 4, and Week 8

SECONDARY OUTCOMES:
Sugar Attachment (HbA1c) | [Time Frame: baseline, 0-4, and 0-8 weeks]
  HbA1C is an indicator of sugar attachment.
Blood Lipids | [Time Frame: baseline, 0-4, and 0-8 weeks].
  Blood lipids are indicators of the body's metabolism and cardiovascular health
Stem cell counts | [Time Frame: baseline, 0-4, and 0-8 weeks]
  Stem cells are indicators of the body's regenerative capacity and biological health
Biomarkers of aging | [Time Frame: baseline, 0-4, and 0-8 weeks]
  Biomarkers of aging are indicators of person's biological age, which may differ from their chronological age, and reflect the rate of aging, health status, and risk of age-related diseases.
Blood Flow Assessment | [Time Frame: baseline, 0-4, and 0-8 weeks]
  Blood flow will be evaluated using the Falcon Quad device, a non-invasive and painless diagnostic tool designed to assess vascular function by measuring and comparing blood pressure across different regions of the body.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Tesla BioHealing Medical Center in Butler-FL, Tampa, Florida
  - Tesla BioHealing Medical Center in Butler-PA, Butler, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data collected during the study, including:
  Demographic data (e.g., age, sex, race/ethnicity)
  Baseline characteristics relevant to the study objectives
  Outcome measures (e.g., clinical scores, response rates, lab values, imaging results)
  Adverse events (frequency, severity, and relationship to the intervention)
  Timepoints of data collection (e.g., baseline, week 1, week 2, follow-up)
  All shared data will be stripped of personally identifiable information in compliance with HIPAA and applicable data privacy regulations.
Supporting Information: Study Protocol, ICF
Time Frame: August 15, 2025, to August 14, 2028
Access Criteria: Access to IPD and Supporting Information:
  Qualified researchers affiliated with academic institutions, healthcare organizations, or regulatory bodies will be able to request access to the individual participant data (IPD) and supporting documents. These documents may include:
  Study protocol
  Statistical analysis plan (SAP)
  Informed consent form (ICF)
  Clinical study report (CSR)
  De-identified IPD, including relevant outcome data
  Access will be granted upon submission and approval of a formal data request outlining the intended use of the data. Researchers will be required to sign a data use agreement (DUA) ensuring the data will be used solely for scientific purposes and that privacy and confidentiality will be maintained.
  Approved users will be provided secure access through a password-protected, encrypted data-sharing platform. No data will be available for download without explicit authorization, and all shared data will comply with applicable data protection regulations.
URL: http://www.firstallmed.org